CLINICAL TRIAL: NCT05835297
Title: Effects of Specifically Developed Exercise on Falls, Physical Functioning, Physical Activity, and General Physical and Psychological Well-being Among Older Adults Dwelling in Nursing Homes Following Recommendations of International Association of Gerontology and Geriatrics-Global Aging Research Network (IAGG-GARN)
Brief Title: Effect of Specifically Developed Exercise Intervention on Falls Among Older Adults in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Munseef Sadaqa, Principal Investigator (PhD candidate), University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9283 - PTE 2022
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-03

CONDITIONS: Fall; Exercise Intervention; Elderly Population
Keywords: Fall; Exercise; Elderly; Guideline; Risk; Functionality
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Physical exercise interventions for 45 min, twice a week plus usual care provided at the nursing home.
  Interventions: Other: Physical exercise interventions
- Usual care (No Intervention): Usual care provided at the nursing home with no specific physical exercise intervention.

INTERVENTIONS:
Other: Physical exercise interventions — Participants will undergo a 12-week multicomponent exercise regimen, twice per week on non-consecutive days for 45-60 min each. The session will be divided into 4 min of warm-up; range of motion exercises of upper and lower extremities, followed by light walking, then 8 min balance exercises, followed by 15 min strength exercises; two sets of 13-15 repetitions maximum of chair rises with progression, two sets of 13-15 repetitions of modified squats (holding a chair backrest if needed) with progression, 2 sets of 20-30 repetitions of seated or 2 sets of 13-15 repetitions of standing calf raises, then 15 min aerobic exercises; five 3-min bouts of walking between two strengthening exercises and/or 2 balance exercises, finally 3 min cool down exercises of light walking and stretching exercises.
  Arms: Exercise group

SUMMARY:
The aim of the study is to examine the effect of multicomponent exercises recommendations on falls, physical functioning, physical activity, and general physical and psychological well-being among Hungarian older adults dwelling in nursing homes.

DETAILED DESCRIPTION:
Methods: Randomized controlled trial of an individually exercise guideline recommended by IAGG-GARN for older males and females living in a nursing home. A stratified randomization will be performed after the baseline assessment. The assessment of primary and secondary outcomes takes place in all subjects upon entry to the study (pre-test) by blinded assessors and at 12 weeks (post-test). After baseline assessments is completed, participants will be randomly allocated to one of the two groups using stratified randomization based on equal distribution of age and gender ratio.

Expected results:

* Reduce the incidence of falls among the nursing homes residents of the intervention group (IG)
* Increase of lower extremity physical functional ability (balance, gait speed, and strength) of the IG
* Improvement of level of physical activity independency of the IG
* Improvement of functional independency of the IG
* Improvement of physical and psychological well-being among IG.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Males and females aged ≥65 years living in nursing homes
* Physically mobile (capable of ambulating/rising from chair with or without assistance)
* Not under simultaneous physical activity/exercise investigation in other experimental studies or under other exercise rehabilitation programme
* To be able to read and understand the self-reported assessments as well as follow the verbal instructions.

Exclusion Criteria:

* Physically unable or medically unfit to participate in physical exercise after consultation of the responsible medical team
* Score of < 18 on mini-mental state examination (MMSE).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of all falls (non-injurious and injurious) | During the 12-week of the intervention.
  Whenever a fall occurred for any of the participants during intervention time, it will be recorded by the staff and reported on a fall incidence report. All fall will be reported; non-injurious (i.e., does not result in a physical harm), moderate injurious falls (i.e., result in bruising, sprains, cuts, abrasions, or reduction in physical function for at least three days, or if the participant sought medical help), and serious injurious falls (i.e., result in a fracture or admission to hospital with an injury or required stitches).

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline and 12th week.
  An instrument to test the lower extremity functionality, it consists of 3 types of balance tests (side-by-side stand, semi-tandem stand, tandem stand), a 4-m gait speed test, and a chair sit-to-stand test. Each domain is scored between 0 and 4 and the overall score ranges from 0 (low mobility/functionality) to 12 (full mobility/ functionality).
Six-minute Walking Test (6MWT) | Baseline and 12th week.
  A timed walk test used to evaluate physical function related to lower extremities strength and mobility. Participants will walk the longest distance possible within 6 min. The outcome is the total walking distance in meters, with higher score indicates better performance.
Timed Up and Go Test (TUGT) | Baseline and 12th week.
  A test to measure functional mobility. The outcome measure will be time in seconds, taken to stand up from a chair, walk 3 m, turn, return to the chair, and sit down. Lower score indicates better performance.
Single Leg Stance Test (SLST) | Baseline and 12th week.
  A test to evaluate the static balance capability. Participants will be asked to stand barefoot on 1leg with eyes open on firm surface for as long as possible; the time in seconds will be recorded using a stopwatch. The participants will complete 3 trials on each leg, and a mean score will be calculated for each leg.
Functional Reach Test (FRT) | Baseline and 12th week.
  A test to evaluate dynamic balance through measuring the maximal distance participants are able to reach forward while standing or sitting on a chair. 3 trials are done and the average of the last two is noted, with longer distance to reach forward indicates better performance.
Mini-mental State Examination (MMSE) | Baseline and 12th week.
  A tool used to evaluate cognitive function (scored from 0 to 30; scores below 24 indicate cognitive impairment) through 11 items.
Barthel Index | Baseline and 12th week.
  A tool is used to record the independence of participants when performing basic activities of daily living (ADLs) via ten items. Feeding, personal toileting, bathing, dressing, and undressing, getting on and off a toilet, controlling bladder, controlling bowel, moving from wheelchair to bed and returning, walking on level surface (or propelling a wheelchair if unable to walk) and ascending and descending stairs are rated on a scale from 0 to 15 points depending on the item. Total possible scores range from 0 (totally dependent) to 100 (fully independent).
World Health Organization Quality of Life questionnaire (WHOQOL-BREF) | Baseline and 12th week.
  A self-administered questionnaire consists of 26 items, evaluating participants' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
World Health Organization Well-Being Index (WHO-5) | Baseline and 12th week.
  A self-reported rating scale of 5 items, measuring subjective psychological well-being.
  The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25.To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Geriatrics Depression Scale (GDS) | Baseline and 12th week.
  A self-rated depression scale of 15 items, that identify symptoms of depression in older adults. A score of ≥ 5 suggests depression.
Beck Depression Inventory (BDI-13) | Baseline and 12th week.
  A 13-question multiple-choice self-report inventory for measuring the severity of depression. A score of ≥ 7 indicates mild depression.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 12th week.
  A self-reported scale for measuring patterns and quality of sleep in adults via 19 items. The global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower score indicates a healthier sleep quality.
Global Physical Activity Questionnaire (GPAQ) | Baseline and 12th week.
  The GPAQ version 2 developed by WHO will be used. It comprises 16 self-administered questions that collect information on physical activity in three settings (or domains) as well as sedentary behaviour of a week (7 days).
Sedentary Behaviour Questionnaire (SBQ) | Baseline and 12th week.
  A self-reported assessment of the amount of time spent doing 9 behaviours separately for weekdays and weekend days. (watching television, playing on a computer/video game, sitting while listening to music, sitting and talking on the phone, doing paperwork or office work, sitting and was reading, playing a musical instrument, doing arts and crafts, sitting and driving/riding in a car, bus, or train).
  Scoring:
  * Convert all times into hours (e.g. a response of 15 minutes or less is recoded as 0.25 and 30 minutes is recoded as 0.5).
  * For total scores of sedentary behavior, sum the hours per day separately for weekday and weekend items.
  * To obtain weekly estimates, weekday hours are multiplied by 5 and weekend hours are multiplied by 2 and these are summed for total hours per week.
  * Estimates over 24 hours per day are truncated to 24 hours per day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Pécs, Hungary

REFERENCES:
- [Derived] Sadaqa M, Debes WA, Nemeth Z, Bera-Baka Z, Vachtler-Szepesi M, Foldes LN, Premusz V, Hock M. Multicomponent exercise intervention for preventing falls and improving physical functioning in older adult nursing home residents: study protocol for a randomised controlled trial. BMC Public Health. 2025 Oct 2;25(1):3296. doi: 10.1186/s12889-025-24606-y. PMID 41039429
- [Derived] Sadaqa M, Debes WA, Nemeth Z, Bera-Baka Z, Vachtler-Szepesi M, Naczine Foldes L, Premusz V, Hock M. Multicomponent Exercise Intervention for Preventing Falls and Improving Physical Functioning in Older Nursing Home Residents: A Single-Blinded Pilot Randomised Controlled Trial. J Clin Med. 2024 Mar 10;13(6):1577. doi: 10.3390/jcm13061577. PMID 38541803